CLINICAL TRIAL: NCT05389540
Title: Overview of Disease Burden in Rural South and Southeast Asia: A Cross-sectional Household Health Survey With Questionnaire Interviews and Selected Laboratory Tests
Brief Title: Rural South and Southeast Asia Household Health Survey
Acronym: SEACTN-HHS
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Mahidol Oxford Tropical Medicine Research Unit (Other); Chiang Rai Clinical Research Unit, Thailand (Unknown); Myanmar Oxford Clinical Research Unit, Yangon, Myanmar (Unknown); Bangladesh Rural Advancement Committee, Dhaka, Bangladesh (Unknown); Cambodia Action for Health Development (AHEAD) (Unknown)
Responsible Party: Sponsor
Other Study IDs: HCR21013
Record Dates: First submitted 2022-05-19; First posted 2022-05-25 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Noncommunicable Disease; Infections; Risk Factors; Health Status
Keywords: Cross-sectional household survey
MeSH Terms: conditions — Noncommunicable Diseases; Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Venous blood samples and Dried blood spot
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- members of selected households at the time of survey: 371 households will be randomly selected from each site in Bangladesh, Cambodia, Myanmar, and Thailand. Assuming each household has an average of 4.5 members and all members will be sampled, 1500 participants will be recruited per site.

SUMMARY:
A cross-sectional household survey with two-stage cluster-randomized sampling. This cross-sectional household survey design to recruit a random sample of households that is representative for each of the study sites. From the selected households, all consenting, household members will be included in the study.

This study is funded by the UK Wellcome Trust. The grant reference number is 215604/Z/19/Z

DETAILED DESCRIPTION:
371 households will be randomly selected from each site in Bangladesh, Cambodia, Myanmar, and Thailand. Assuming each household has an average of 4.5 members and all members will be sampled, 1500 participants will be recruited per site. This sample size allows for the overall prevalence estimation of key survey indicators with 95% confidence and 5% degree of precision.

The survey components include questionnaire interview, physical examination, blood sample collection, and point of care (PoC) tests. The questionnaire interview will collect information on household characteristics, members' disability, presence or history of disease, risk factors, self-perceived quality of life, and health seeking behaviour. For women, questions about reproductive health and antenatal care, and for young children, vaccination coverage and achievement of child development goals, will also be assessed.

For physical examinations, tympanic temperature, weight and height will be measured in all household members, mid-upper arm circumference in young children, and blood pressure in adults. Blood sample will be collected from all participants aged 6 months and above. Venous blood samples will be collected from participants aged 5 years and older, and dried blood spot will be collected from children under 5 years. Samples will be shipped to a central laboratory and analysed. Haemoglobin PoC will be administered to all participants.

All data will be collected directly on an electronic case report form using tablets, and uploaded to an electronic database.

ELIGIBILITY:
Inclusion Criteria:

* All members of the selected households at the time of the survey; and able to provide informed consent.

Exclusion Criteria:

* Adults or children whose parent/guardian/ caretaker are unable or unwilling to provide informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Households located in the survey villages and identified in the household list are eligible for the survey. All members of the randomly selected households will be recruited
Sampling Method: Probability Sample
Enrollment: 4747 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of long-lasting antibodies (IgG) against selected causes of non-malaria febrile illnesses | Upon enrollment
Prevalence of Plasmodium spp. by PCR | Upon enrollment
Prevalence of chronic Hepatitis B and C | Upon enrollment
Prevalence of selected non-communicable diseases (e.g. diabetes, chronic obstructive pulmonary diseases, stroke) according to self-reported disease history and laboratory tests | Upon enrollment
Prevalence of reported disability | Upon enrollment
Lifetime prevalence of reported injury or death caused by an accident | Upon enrollment
Self-rated overall health status | Upon enrollment
Questionnaire evaluation of health-related quality of life | Upon enrollment
Prevalence of self-reported tobacco, alcohol, and other substitute use among the population aged 15 and above | Upon enrollment
Prevalence of underweight and overweight, raised blood pressure and total cholesterol | Upon enrollment

SECONDARY OUTCOMES:
Evaluation of household wealth quartile according to self-reported household characteristics | Upon enrollment
Education level, marital status, and occupation | Upon enrollment
Self-reported health-related household characteristics (e.g. household cooking fuel, source of drinking water, possession of mosquito net) | Upon enrollment
Proportion of population self-reported having sought for medical care in the past month, and care providers visited | Upon enrollment
Self-reported antenatal care coverage among women who have ever given birth | Upon enrollment
Reported vaccination coverage among children < 3 years | Upon enrollment
Prevalence of reported exclusive breast feeding among children < 5 years | Upon enrollment
Prevalence of children aged 3-4 years who have reached early child development milestones, reported by caretaker | Upon enrollment
Presence of self-reported symptoms or diagnosed illness besides the outcome measures of the primary objectives | Upon enrollment
Reported illness in the last month and type of illness | Upon enrollment
Prevalence of IgM antibodies against selected acute non-malaria causes of febrile illness | Upon enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Yoel Lubell, Professor, Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit; Thomas Peto, PhD, Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit
Locations (4):
- BangladeshBuilding Resources Across Communities (BRAC), Dhaka, Bangladesh
- Medical Action Myanmar (MAM), Yangon, Burma
- Cambodia Action for Health Development (AHEAD), Battambang, Cambodia
- Chiangrai Clinical Research Unit (CCRU), Chiang Rai, Thailand

IPD SHARING:
Plan to Share IPD: Yes
With participant's consent, clinical data and results from blood analyses stored in the database may be shared according to the terms defined in the MORU data sharing policy with other researchers to use in the future.
Time Frame: After completion of survey activities and reporting
Access Criteria: MORU Data Sharing Policy
URL: https://www.tropmedres.ac/units/moru-bangkok/bioethics-engagement/data-sharing/moru-tropical-network-policy-on-sharing-data-and-other-outputs

REFERENCES:
- [Background] Chandna A, Chew R, Shwe Nwe Htun N, Peto TJ, Zhang M, Liverani M, Brummaier T, Phommasone K, Perrone C, Pyae Phyo A, Sattabongkot J, Roobsoong W, Nguitragool W, Sen A, Ibna Zaman S, Sandar Zaw A, Batty E, Waithira N, Abdad MY, Blacksell SD, Bodhidatta L, Callery JJ, Fagnark W, Huangsuranun W, Islam S, Lertcharoenchoke S, Lohavittayavikant S, Mukaka M, Moul V, Kumer Neogi A, Nedsuwan S, Pongvongsa T, Ponsap P, Richard-Greenblatt M, Schilling WHK, Thaipadungpanit J, Tripura R, Dondorp AM, Mayxay M, White NJ, Nosten F, Smithuis F, Ashley EA, Maude RJ, Day NPJ, Lubell Y. Defining the burden of febrile illness in rural South and Southeast Asia: an open letter to announce the launch of the Rural Febrile Illness project. Wellcome Open Res. 2022 Mar 10;6:64. doi: 10.12688/wellcomeopenres.16393.2. eCollection 2021. PMID 34017924
- [Derived] Zhang M, Htun NSN, Islam S, Sen A, Islam A, Neogi AK, Tripura R, Dysoley L, Perrone C, Chew R, Batty EM, Thongpiam W, Wongsantichon J, Menggred C, Zaman SI, Waithira N, Blacksell S, Liverani M, Lee S, Maude RJ, Day NPJ, Lubell Y, Peto TJ. Defining the hidden burden of disease in rural communities in Bangladesh, Cambodia and Thailand: a cross-sectional household health survey protocol. BMJ Open. 2024 Mar 23;14(3):e081079. doi: 10.1136/bmjopen-2023-081079. PMID 38521526
- See also: Related Info — https://seactn.org/